CLINICAL TRIAL: NCT04989647
Title: An International Randomised Trial of Radical Surgery Followed by Adjuvant (Chemo)Radiation Versus no Further Treatment in Patients With Early-stage, Intermediate-risk Cervical Cancer Patients
Brief Title: Intermediate Risk Cervical Cancer: Radical Surgery +/- Adjuvant Radiotherapy
Acronym: CERVANTES
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The Central and Eastern European Gynecologic Oncology Group (Other)
Responsible Party: Principal Investigator, David Cibula, prof. David Cibula, MD, PhD, General University Hospital, Prague
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ENGOT-cx16/CEEGOG/CERVANTES
Record Dates: First submitted 2021-07-29; First posted 2021-08-04 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Cervical Cancer
Keywords: intermediate risk cervical cancer; adjuvant radiotherapy; disease free survival
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Radiotherapy, Adjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A: Surgery only (Experimental): Radical hysterectomy, sentinel lymph node biopsy and systematic pelvic lymphadenectomy (PLND)*. No further treatment will be administered.
  *PLND can be avoided in patients with tumours < 4cm
  Interventions: Radiation: No adjuvant therapy
- B: Surgery + radiothrerapy (Experimental): Radical hysterectomy, sentinel lymph node biopsy and systematic pelvic lymphadenectomy (PLND)*, followed by adjuvant treatment.
  *PLND can be avoided in patients with tumours < 4cm
  Interventions: Radiation: Adjuvant radiotherapy

INTERVENTIONS:
Radiation: No adjuvant therapy — Patients will not receive any type of adjuvant therapy.
  Arms: A: Surgery only
Radiation: Adjuvant radiotherapy — Patients will receive adjuvant treatment composed of either pelvic radiotherapy external beam radiotherapy ± brachytherapy or concomitant chemoradiotherapy (pelvic radiotherapy + chemotherapy).
  Arms: B: Surgery + radiothrerapy

SUMMARY:
The objective of the trial is to evaluate if adjuvant (chemo)radiation is associated with a disease-free survival benefit after radical surgery in patients with intermediate risk cervical cancer. The primary endpoint of the study is the disease-free survival from the day of randomisation. A total of 514 patients are required to achieve 80% power on 5% significance level with non-inferiority margin of 5% to test the difference between the ARMs using Cox proportional hazards model. The maximal tolerated margin for non-inferiority in 2-year DFS is 5% (including expected drop-out rate of 10%).

DETAILED DESCRIPTION:
The role of adjuvant (chemo)radiotherapy in intermediate risk (IR) cervical cancer patients is controversial, supported by single randomised GOG 92 study performed more than 20 years ago. Intermediate-risk group is defined as lymph node negative but with a combination of negative prognostic factors (tumour size >2 cm, lymphovascular space invasion, deep stromal invasion >2/3). Recent retrospective studies showed excellent local control in intermediate risk group patients after radical surgery with no additional adjuvant treatment.

CERVANTES trial is designed to bring level A evidence on the role of adjuvant treatment in IR patients in an international, prospective, randomised study. Patients will be registered into the trial before surgery and randomised after the final pathology report has been received into ARM A, with no additional treatment, and ARM B, receiving adjuvant (chemo)radiotherapy. Quality assurance program will be in place for both, radical surgery and adjuvant treatment.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed invasive cervical cancer
* FIGO IB1-IIA
* Squamous cell cancer or HPV-related adenocarcinoma
* Presence of tumour-related risk factors as follows:

  1. tumour ≥4 cm OR
  2. tumour>2 cm <4 cm AND lymphovascular space invasion OR
  3. tumour >2 cm <4 cm AND tumour free distance <3 mm OR
  4. tumour >2 cm <4 cm AND deep stromal invasion (>2/3)
* No evidence of suspicious pelvic lymph nodes or distant metastases on imaging (by radiological subjective assessment before surgery and negative pelvic LN on final pathology)
* ECOG performance status 0-1
* Deemed suitable and fit for radical surgery followed by adjuvant radiotherapy
* Negative pregnancy test (if applicable)
* Negative HIV test (only performed in high-risk countries or patients who have moved from those countries within the past 10 years)

Exclusion Criteria:

* Adenosquamous cancer or adenocarcinoma unusual type (non-HPV related - such as: mucinous, clear cell, mesonephric) or other rare tumour types (those not listed in the inclusion criteria)
* Inconclusive primary site of disease
* Unequivocally positive lymph node by imaging (by radiological subjective assessment)
* FIGO <IB1 / >IIA
* Previous pelvic malignancy
* History of second primary cancer outside pelvis if ≤ 3 years complete clinical remission (CCR)
* Previous pelvic radiotherapy
* Neoadjuvant chemotherapy prior surgical treatment
* Low likelihood of patient compliance to the follow-up

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 514 (Estimated)
Dates: Start 2022-06-10 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | Analysed 3 years after randomization of the last patient.
  Calculated as an interval from the day of randomisation until diagnosis of recurrence: (a) unequivocal finding on imaging by subjective radiological assessment; b) suspicious recurrence on imaging either confirmed by biopsy or supported by other signs (disease progression on imaging or progression of symptoms); (c) physical examination supported by clinical evidence (i.e., symptoms or progression); or (d) death caused by disease or death of unknown cause.

SECONDARY OUTCOMES:
Overall survival | Analysed 6 years after randomization of the last patient.
Pelvic disease-free survival | Analysed 3 years after randomization of the last patient.
Health-related quality of life based questionnaire | Analysed 3 years after randomization of the last patient.
  The analysis will be made based on EORTC validated questionnaires and developed qualitative CERVANTES questionnaire.
Treatment-related adverse events based on Common Terminology Criteria for Adverse Events v5.0 | Analysed 3 years after randomization of the last patient.

CONTACTS AND LOCATIONS:
Overall Officials: David Cibula, prof., Principal Investigator — General University Hospital in Prague, Czech Republic
Locations (1):
- General University Hospital in Prague, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sedlis A, Bundy BN, Rotman MZ, Lentz SS, Muderspach LI, Zaino RJ. A randomized trial of pelvic radiation therapy versus no further therapy in selected patients with stage IB carcinoma of the cervix after radical hysterectomy and pelvic lymphadenectomy: A Gynecologic Oncology Group Study. Gynecol Oncol. 1999 May;73(2):177-83. doi: 10.1006/gyno.1999.5387. PMID 10329031
- [Background] Rotman M, Sedlis A, Piedmonte MR, Bundy B, Lentz SS, Muderspach LI, Zaino RJ. A phase III randomized trial of postoperative pelvic irradiation in Stage IB cervical carcinoma with poor prognostic features: follow-up of a gynecologic oncology group study. Int J Radiat Oncol Biol Phys. 2006 May 1;65(1):169-76. doi: 10.1016/j.ijrobp.2005.10.019. Epub 2006 Jan 19. PMID 16427212
- [Background] Scharl S, Becher C, Gerken M, Scharl A, Anapolski M, Ignatov A, Inwald EC, Ortmann O, Kolbl O, Klinkhammer-Schalke M, Papathemelis T. Is there a benefit for adjuvant radio(chemo)therapy in early cervical cancer? Results from a population-based study. Arch Gynecol Obstet. 2021 Sep;304(3):759-771. doi: 10.1007/s00404-021-05989-w. Epub 2021 Feb 11. PMID 33575846
- [Background] Kim SI, Kim TH, Lee M, Kim HS, Chung HH, Lee TS, Jeon HW, Kim JW, Park NH, Song YS. Impact of Adjuvant Radiotherapy on Survival Outcomes in Intermediate-Risk, Early-Stage Cervical Cancer: Analyses Regarding Surgical Approach of Radical Hysterectomy. J Clin Med. 2020 Nov 3;9(11):3545. doi: 10.3390/jcm9113545. PMID 33153125
- [Background] Cibula D, Abu-Rustum NR, Fischerova D, Pather S, Lavigne K, Slama J, Alektiar K, Ming-Yin L, Kocian R, Germanova A, Fruhauf F, Dostalek L, Dusek L, Narayan K. Surgical treatment of "intermediate risk" lymph node negative cervical cancer patients without adjuvant radiotherapy-A retrospective cohort study and review of the literature. Gynecol Oncol. 2018 Dec;151(3):438-443. doi: 10.1016/j.ygyno.2018.10.018. Epub 2018 Oct 20. PMID 30348519
- [Background] van der Velden J, Mom CH, van Lonkhuijzen L, Tjiong MY, Westerveld H, Fons G. Analysis of isolated loco-regional recurrence rate in intermediate risk early cervical cancer after a type C2 radical hysterectomy without adjuvant radiotherapy. Int J Gynecol Cancer. 2019 Jun 2;29(5):874-878. doi: 10.1136/ijgc-2019-000445. PMID 31133601
- [Background] Cao L, Wen H, Feng Z, Han X, Zhu J, Wu X. Role of adjuvant therapy after radical hysterectomy in intermediate-risk, early-stage cervical cancer. Int J Gynecol Cancer. 2021 Jan;31(1):52-58. doi: 10.1136/ijgc-2020-001974. Epub 2020 Dec 10. PMID 33303568
- [Background] Akilli H, Tohma YA, Bulut AN, Karakas LA, Haberal AN, Kuscu UE, Ayhan A. Comparison of no adjuvant treatment and radiotherapy in early-stage cervical carcinoma with intermediate risk factors. Int J Gynaecol Obstet. 2020 Jun;149(3):298-302. doi: 10.1002/ijgo.13147. Epub 2020 Apr 22. PMID 32246761
- [Background] Nasioudis D, Latif NA, Giuntoli Ii RL, Haggerty AF, Cory L, Kim SH, Morgan MA, Ko EM. Role of adjuvant radiation therapy after radical hysterectomy in patients with stage IB cervical carcinoma and intermediate risk factors. Int J Gynecol Cancer. 2021 Jun;31(6):829-834. doi: 10.1136/ijgc-2021-002489. Epub 2021 May 6. PMID 33962994
- [Background] Rogers L, Siu SS, Luesley D, Bryant A, Dickinson HO. Radiotherapy and chemoradiation after surgery for early cervical cancer. Cochrane Database Syst Rev. 2012 May 16;2012(5):CD007583. doi: 10.1002/14651858.CD007583.pub3. PMID 22592722
- [Background] Bilek K, Ebeling K, Leitsmann H, Seidel G. Radical pelvic surgery versus radical surgery plus radiotherapy for stage Ib carcinoma of the cervix uteri. Preliminary results of a prospective randomized clinical study. Arch Geschwulstforsch. 1982 May;52(3):223-9. PMID 6751268
- [Background] Schorge JO, Molpus KL, Koelliker D, Nikrui N, Goodman A, Fuller AF Jr. Stage IB and IIA cervical cancer with negative lymph nodes: the role of adjuvant radiotherapy after radical hysterectomy. Gynecol Oncol. 1997 Jul;66(1):31-5. doi: 10.1006/gyno.1997.4691. PMID 9234917
- [Background] Kridelka FJ, Berg DO, Neuman M, Edwards LS, Robertson G, Grant PT, Hacker NF. Adjuvant small field pelvic radiation for patients with high risk, stage IB lymph node negative cervix carcinoma after radical hysterectomy and pelvic lymph node dissection. A pilot study. Cancer. 1999 Nov 15;86(10):2059-65. PMID 10570432
- [Background] Hong JH, Tsai CS, Lai CH, Chang TC, Wang CC, Lee SP, Tseng CJ, Hsueh S. Postoperative low-pelvic irradiation for stage I-IIA cervical cancer patients with risk factors other than pelvic lymph node metastasis. Int J Radiat Oncol Biol Phys. 2002 Aug 1;53(5):1284-90. doi: 10.1016/s0360-3016(02)02831-6. PMID 12128131
- [Background] Pieterse QD, Trimbos JB, Dijkman A, Creutzberg CL, Gaarenstroom KN, Peters AA, Kenter GG. Postoperative radiation therapy improves prognosis in patients with adverse risk factors in localized, early-stage cervical cancer: a retrospective comparative study. Int J Gynecol Cancer. 2006 May-Jun;16(3):1112-8. doi: 10.1111/j.1525-1438.2006.00600.x. PMID 16803494
- [Background] Chen SW, Liang JA, Yang SN, Lin FJ. Early stage cervical cancer with negative pelvic lymph nodes: pattern of failure and complication following radical hysterectomy and adjuvant radiotherapy. Eur J Gynaecol Oncol. 2004;25(1):81-6. PMID 15053068
- [Background] Cibula D, Slama J, Dostalek L, Fischerova D, Germanova A, Fruhauf F, Dundr P, Nemejcova K, Jarkovsky J, Sebestova S, Burgetova A, Borcinova M, Kocian R. Tumour-free distance: a novel prognostic marker in patients with early-stage cervical cancer treated by primary surgery. Br J Cancer. 2021 Mar;124(6):1121-1129. doi: 10.1038/s41416-020-01204-w. Epub 2020 Dec 14. PMID 33318656
- [Background] Cibula D, Potter R, Planchamp F, Avall-Lundqvist E, Fischerova D, Haie Meder C, Kohler C, Landoni F, Lax S, Lindegaard JC, Mahantshetty U, Mathevet P, McCluggage WG, McCormack M, Naik R, Nout R, Pignata S, Ponce J, Querleu D, Raspagliesi F, Rodolakis A, Tamussino K, Wimberger P, Raspollini MR. The European Society of Gynaecological Oncology/European Society for Radiotherapy and Oncology/European Society of Pathology guidelines for the management of patients with cervical cancer. Radiother Oncol. 2018 Jun;127(3):404-416. doi: 10.1016/j.radonc.2018.03.003. Epub 2018 May 1. PMID 29728273
- [Derived] Cibula D, Borcinova M, Kocian R, Feltl D, Argalacsova S, Dvorak P, Fischerova D, Dundr P, Jarkovsky J, Hoschlova E, Slama J, Scambia G. CERVANTES: an international randomized trial of radical surgery followed by adjuvant (chemo) radiation versus no further treatment in patients with early-stage, intermediate-risk cervical cancer (CEEGOG-CX-05; ENGOT-CX16). Int J Gynecol Cancer. 2022 Oct 3;32(10):1327-1331. doi: 10.1136/ijgc-2022-003918. PMID 36100282